CLINICAL TRIAL: NCT03253835
Title: Cardiac Blood Flow Patterns Associated With Regional and Global Left Ventricular Myocardial Damage: an Explorative Study by Cardiac Magnetic Resonance
Brief Title: Cardiac Blood Flow Patterns Associated With Left Ventricular Myocardial Damage
Acronym: CMR-LHD
Status: Enrolling by invitation | Type: Observational
Sponsor: Medical University of Graz (Other)
Collaborators: Anniversary Fund of the Oesterreichische Nationalbank (Unknown)
Responsible Party: Principal Investigator, Ursula Reiter, PD DI Dr., Medical University of Graz
Other Study IDs: CMR-12-LHD
Record Dates: First submitted 2017-08-16; First posted 2017-08-18 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Cardiomyopathies; Myocardial Injury; Healthy
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Myocardial Injury: patients with myocardial injuries due to ischemic heart disease, patients with myocardial injuries due to non-ischemic heart disease.
  Interventions: Diagnostic Test: Single Group Assignment
- No Myocardial Injury: subjects without myocardial injuries with normal cardiac function subjects without myocardial injuries with altered cardiac function
  Interventions: Diagnostic Test: Single Group Assignment

INTERVENTIONS:
Diagnostic Test: Single Group Assignment

SUMMARY:
Various factors affect the performance of the heart: The contractile properties of myocardial muscle cells are the fundamental devices for translating tension-generation and shortening of the cardiac muscle into pressure-generation and blood volume ejection from the heart into the body. On the other hand, the performance of heart can be analyzed with respect to input and output of blood to/from the hollow cardiac muscle and evaluated in terms of the performance of a pump: With every heartbeat blood is sucked from a low-pressure system (veins) and pumped to the arterial high-pressure system via one-way valves, whereas efficiency, ejected blood volume, blood flow and pressures are linked by hemodynamic laws.

Cardiac magnetic resonance (CMR) is the "gold standard technique" to determine cardiac function and muscle mass, as well as for non-invasive diagnosis of myocardial necrosis/fibrosis. Furthermore, new CMR imaging techniques enabling the measurement of myocardial magnetic relaxation times for characterization of myocardial morphology and the acquisition of time-resolved, three-dimensional blood flow velocity fields in the heart and surrounding vessels, represent promising tools for the evaluation of the interaction between myocardial morphology and cardiac function.

Aim of this explorative study is to 1. identify myocardial pathology-associated blood flow patterns in the heart and surrounding great vessels, and 2. correlate characteristic blood flow patterns in the heat (existence of vortices, vorticity, vortex formation, propagation dynamics …) with myocardial injuries.

ELIGIBILITY:
Inclusion Criteria:

* patients age 20-80 years,
* patients with and without ischemic or non-ischemic myocardial injuries scheduled for routine cardiac magnetic resonance imaging,
* ability to hold the breath,
* ability to give informed consent

Exclusion Criteria:

* patients with metal devices or other magnetic material in or on the subjects body which will be hazardous for magnetic resonance investigation (e.g. heart pace-maker, brain aneurysm clip, nerve stimulators, electrodes, penile implants, colored contact lenses, patch to deliver medications through the skin, any metal implants as rods, joints, plates, pins, screws, nails or clips, embolization coil, or any metal fragments or shrapnel in the body),
* patients with tendency toward claustrophobia,
* hemodynamically unstable patients,
* patients with (major) arrhythmia
* pregnancy,
* impaired kidney function indicated by creatin clearance lower than 60 ml/min (creatin clearance will be calculated according to Cockroft-Gault formula)

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients referred to CMR investigation. If suitable and inclusion criteria are met, the patient will be asked if she/he is interested in participating in this study. Participation means, that aside from the respective routine CMR protocol, additional images will be taken within the investigation resulting in 15-20 minutes extra investigation time.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2013-11-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Myocardial pathology-associated blood flow patterns in the heart and surrounding great vessels | 2 years
  Morphologic, functional and blood flow CMR parameters will be evaluated with different techniques. Cardiac blood flow pattern parameters will be correlated with myocardial injury derived non-invasively from late gadolinium enhancement

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fuchsjäger, Univ.-Prof., Study Chair — Medical Universtiy of Graz; Ursula Reiter, PD DI Dr., Principal Investigator — Medical Universtiy of Graz
Locations (1):
- Medical Unitersity Graz, Department of Radiology, Division of General Radiology, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Krauter C, Reiter U, Reiter C, Nizhnikava V, Schmidt A, Stollberger R, Fuchsjager M, Reiter G. Impact of the Choice of Native T1 in Pixelwise Myocardial Blood Flow Quantification. J Magn Reson Imaging. 2021 Mar;53(3):755-765. doi: 10.1002/jmri.27375. Epub 2020 Oct 8. PMID 33034120
- [Result] Krauter C, Reiter U, Reiter C, Nizhnikava V, Masana M, Schmidt A, Fuchsjager M, Stollberger R, Reiter G. Automated mitral valve vortex ring extraction from 4D-flow MRI. Magn Reson Med. 2020 Dec;84(6):3396-3408. doi: 10.1002/mrm.28361. Epub 2020 Jun 18. PMID 32557819
- [Result] Reiter C, Reiter G, Krauter C, Kolesnik E, Greiser A, Scherr D, Schmidt A, Fuchsjager M, Reiter U. Impact of the evaluation method on 4D flow-derived diastolic transmitral and myocardial peak velocities: Comparison with echocardiography. Eur J Radiol. 2024 Jan;170:111247. doi: 10.1016/j.ejrad.2023.111247. Epub 2023 Dec 5. PMID 38071909